CLINICAL TRIAL: NCT02640157
Title: A Randomized, Open-Label, Active-Controlled, Multicenter Study to Compare Efficacy and Safety of ABT-493/ABT-530 to Sofosbuvir Co-Administered With Daclatasvir in Adults With Chronic Hepatitis C Virus Genotype 3 Infection (ENDURANCE-3)
Brief Title: A Study Comparing Efficacy and Safety of ABT-493/ABT-530 to Sofosbuvir Dosed With Daclatasvir in Adults With HCV Genotype 3 Infection
Acronym: ENDURANCE-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-594; 2015-002272-24 (EudraCT Number)
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus; Genotype 3 Hepatitis C Virus
Keywords: interferon free; Hepatitis C; daclatasvir; Sovaldi; HCV; Hepatitis C Virus; Hepatitis C Genotype 3; Hep C; sofosbuvir; Chronic Hepatitis C; Daklinza
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir; Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 12 weeks.
  Interventions: Drug: ABT-493/ABT-530
- Arm B (Active Comparator): Sofosbuvir 400 mg once daily (QD) co-administered with daclatasvir 60 mg QD for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir
- Arm C (Experimental): ABT-493/ABT-530 (300 mg/120 mg) coformulated once daily (QD) for 8 weeks.
  Interventions: Drug: ABT-493/ABT-530

INTERVENTIONS:
Drug: ABT-493/ABT-530 — Tablet; ABT-493 coformulated with ABT-530
  Other Names: ABT-493 also known as glecaprevir; ABT-530 also known as pibrentasvir; MAVYRET
  Arms: Arm A; Arm C
Drug: Sofosbuvir — Tablet
  Other Names: Sovaldi
  Arms: Arm B
Drug: Daclatasvir — Tablet
  Other Names: Daklinza
  Arms: Arm B

SUMMARY:
The purpose of this study was to compare the safety and efficacy of ABT-493/ABT-530 to the combination of sofosbuvir (SOF) and daclatasvir (DCV) in adults with genotype 3 (GT3) chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This study was a Phase 3, randomized, open-label, active-controlled multicenter study to compare efficacy and safety of ABT-493/ABT-530 to SOF and DCV in treatment-naïve chronic HCV GT3-infected participants without cirrhosis. The study consisted of 2 periods, a treatment period (participants received 8 or 12 weeks of ABT-493/ABT-530 or 12 weeks of SOF with DCV) and a post-treatment period (participants who completed or prematurely discontinued the treatment period were followed for 24 weeks after their last dose of study drug to evaluate efficacy and to monitor HCV RNA and the emergence and persistence of viral variants).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of nonchildbearing potential, practicing total abstinence, sexually active with female partners only, or using allowed contraceptive methods) at least 18 years of age at time of screening.
* Screening laboratory result indicating HCV GT3 infection.
* Chronic HCV infection, defined as one of the following:

  * Positive for anti-HCV antibody (Ab) or HCV RNA at least 6 months before screening; or
  * A liver biopsy consistent with chronic HCV infection; or
  * Abnormal alanine aminotransferase (ALT) levels for at least 6 months before screening.
* Hepatitis C virus treatment-naïve (i.e., participant had never received any anti-HCV treatment).
* Documented as noncirrhotic.

Exclusion Criteria:

* Female who was pregnant, planning to become pregnant during the study, or breastfeeding; or male whose partner was pregnant or planning to become pregnant during the study.
* Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse that could have precluded adherence to the protocol in the opinion of the investigator.
* Positive test result at screening for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus Ab (HIV Ab).
* Hepatitis C virus genotyping performed during screening indicated co-infection with more than one HCV genotype.
* Any cause of liver disease other than chronic HCV infection.
* Consideration by the investigator, for any reason, that the participant was an unsuitable candidate to receive ABT-493/ABT-530, SOF, or DCV.
* History of severe, life-threatening, or other significant sensitivity to any excipients of the study drug.
* Previous use of any anti-HCV treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeuzem S, Foster GR, Wang S, Asatryan A, Gane E, Feld JJ, Asselah T, Bourliere M, Ruane PJ, Wedemeyer H, Pol S, Flisiak R, Poordad F, Chuang WL, Stedman CA, Flamm S, Kwo P, Dore GJ, Sepulveda-Arzola G, Roberts SK, Soto-Malave R, Kaita K, Puoti M, Vierling J, Tam E, Vargas HE, Bruck R, Fuster F, Paik SW, Felizarta F, Kort J, Fu B, Liu R, Ng TI, Pilot-Matias T, Lin CW, Trinh R, Mensa FJ. Glecaprevir-Pibrentasvir for 8 or 12 Weeks in HCV Genotype 1 or 3 Infection. N Engl J Med. 2018 Jan 25;378(4):354-369. doi: 10.1056/NEJMoa1702417. PMID 29365309
- [Derived] Brown A, Welzel TM, Conway B, Negro F, Brau N, Grebely J, Puoti M, Aghemo A, Kleine H, Pugatch D, Mensa FJ, Chen YJ, Lei Y, Lawitz E, Asselah T. Adherence to pan-genotypic glecaprevir/pibrentasvir and efficacy in HCV-infected patients: A pooled analysis of clinical trials. Liver Int. 2020 Apr;40(4):778-786. doi: 10.1111/liv.14266. Epub 2019 Oct 18. PMID 31568620
- [Derived] Back D, Belperio P, Bondin M, Negro F, Talal AH, Park C, Zhang Z, Pinsky B, Crown E, Mensa FJ, Marra F. Efficacy and safety of glecaprevir/pibrentasvir in patients with chronic HCV infection and psychiatric disorders: An integrated analysis. J Viral Hepat. 2019 Aug;26(8):951-960. doi: 10.1111/jvh.13110. Epub 2019 May 20. PMID 30977945
- [Derived] Gane E, Poordad F, Zadeikis N, Valdes J, Lin CW, Liu W, Asatryan A, Wang S, Stedman C, Greenbloom S, Nguyen T, Elkhashab M, Worns MA, Tran A, Mulkay JP, Setze C, Yu Y, Pilot-Matias T, Porcalla A, Mensa FJ. Safety and Pharmacokinetics of Glecaprevir/Pibrentasvir in Adults With Chronic Genotype 1-6 Hepatitis C Virus Infections and Compensated Liver Disease. Clin Infect Dis. 2019 Oct 30;69(10):1657-1664. doi: 10.1093/cid/ciz022. PMID 30923816
- [Derived] Foster GR, Dore GJ, Wang S, Grebely J, Sherman KE, Baumgarten A, Conway B, Jackson D, Asselah T, Gschwantler M, Tomasiewicz K, Aguilar H, Asatryan A, Hu Y, Mensa FJ. Glecaprevir/pibrentasvir in patients with chronic HCV and recent drug use: An integrated analysis of 7 phase III studies. Drug Alcohol Depend. 2019 Jan 1;194:487-494. doi: 10.1016/j.drugalcdep.2018.11.007. Epub 2018 Nov 24. PMID 30529905
- [Derived] Flamm S, Reddy KR, Zadeikis N, Hassanein T, Bacon BR, Maieron A, Zeuzem S, Bourliere M, Calleja JL, Kosloski MP, Oberoi RK, Lin CW, Yu Y, Lovell S, Semizarov D, Mensa FJ. Efficacy and Pharmacokinetics of Glecaprevir and Pibrentasvir With Concurrent Use of Acid-Reducing Agents in Patients With Chronic HCV Infection. Clin Gastroenterol Hepatol. 2019 Feb;17(3):527-535.e6. doi: 10.1016/j.cgh.2018.07.003. Epub 2018 Sep 10. PMID 30012435
- See also: Related info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 506 participants were randomized and 505 received ≥ 1 dose of study drug. One participant in Arm B was randomized in error and never dispensed study drug. This participant is included in the total number of participants in Arm B who discontinued the study. This study included a 42-day screening period.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 233 (Intent-to-treat population: all participants who received at least 1 dose of study drug) | 116 | 157 (Intent-to-treat population: all participants who received at least 1 dose of study drug)
Received Study Drug | 233 | 115 (One participant in Arm B was randomized in error and never dispensed study drug.) | 157
Completed Study Drug | 225 | 112 | 154
Discontinued Study Drug | 8 | 3 | 3
Completed | 220 | 111 | 147
Not Completed | 13 | 5 | 10
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Withdrew consent | 2 | 0 | 2
Not completed — Lost to Follow-up | 9 | 2 | 7
Not completed — Randomized in error; did not receive Tx | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug (safety population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 233 | 115 | 157 | 505
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.18 (10.68) | 47.06 (11.31) | 45.43 (12.19) | 46.61 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 63 | 64 | 239
  Male | 121 | 52 | 93 | 266

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12): Noninferiority of Arm A to Arm B
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ] 12 weeks after the last dose of study drug. The primary efficacy endpoint was noninferiority in the percentage of participants achieving SVR12 of the 12-week regimen (Arm A) to the standard of care (Arm B: 12 weeks of treatment with sofosbuvir [SOF] + daclatasvir [DCV]), defined as: a) the lower bound of the 95% confidence interval (CI) for the difference was above the non-inferiority margin of -6% and the lower bound of the 95% CI for the SVR12 rate within Arm A was greater than 92%; OR b) the lower bound of the 95% CI for the difference was below the non-inferiority margin of -6% and the lower bound of the 97.5% CI for the SVR12 rate within Arm A was greater than 92%; OR c) the lower bound of the 97.5% CI for the difference was above the non-inferiority margin of -6% and the lower bound of the 95% CI for the SVR12 rate within Arm A was below 92%.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat population: all participants who received at least 1 dose of study drug; participants with missing data after backwards imputation were counted as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 233 | 115
percentage of participants | 95.3 [92.6 to 98.0] | 96.5 [93.2 to 99.9]
Statistical Analysis 1: Comparison: Arm A vs Arm B; Difference in SVR12 rates (Arm A - Arm B); Test type: Non-Inferiority — Noninferiority: a) the lower bound (LB) of the 95%CI for the difference was above the non-inferiority margin of -6% and the LB of the 95%CI for the SVR12 rate within Arm A was >92%; or b) the LB of the 95%CI for the difference was below the non-inferiority margin of -6% and the LB of the 97.5%CI for the SVR12 rate within Arm A was >92%; or c) the LB of the 97.5%CI for the difference was above the non-inferiority margin of -6% and the LB of the 95%CI for the SVR12 rate within Arm A was below 92%; Difference in percentage of participants = -1.2, 95% CI 2-sided [-5.6 to 3.1]
Statistical Analysis 2: Comparison: Arm A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; percentage of participants = 95.3, 97.5% CI 2-sided [92.2 to 98.4]
Statistical Analysis 3: Comparison: Arm A vs Arm B; Difference in SVR12 rates (Arm A - Arm B); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentage of participants = -1.2, 97.5% CI 2-sided [-6.2 to 3.7]

2. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12): Noninferiority of Arm C to Arm A
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug. If the first primary efficacy objective (noninferiority of Arm A to Arm B) was achieved, then the second primary efficacy objective, noninferiority in the percentage of participants achieving SVR12 of the 8-week regimen (Arm C) to the 12-week regimen (Arm A) was to be tested. Noninferiority was defined as: a) the lower bound of the 95% CI for the difference was above the noninferiority margin of -6% and the lower bound of the 95% CI for the SVR12 rate within Arm C was greater than 92%, OR b) the lower bound of the 95% CI for the difference was below the noninferiority margin of -6% and the lower bound of the 97.5% CI for the SVR12 rate within Arm C was greater than 92%, OR c) the lower bound of the 97.5% CI for the difference was above the noninferiority margin of -6% and the lower bound of the 95% CI for the SVR12 rate within Arm C was below 92%.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population); participants with missing data after backwards imputation were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm C
Number analyzed (Participants) | 233 | 157
percentage of participants | 95.3 [92.6 to 98.0] | 94.9 [91.5 to 98.3]
Statistical Analysis 1: Comparison: Arm A vs Arm C; Difference in SVR12 rates (Arm C - Arm A); Test type: Non-Inferiority — Noninferiority: a) the lower bound (LB) of the 95%CI for the difference was above the non-inferiority margin of -6% and the LB of the 95%CI for the SVR12 rate within Arm C was >92%; or b) the LB of the 95%CI for the difference was below the non-inferiority margin of -6% and the LB of the 97.5%CI for the SVR12 rate within Arm C was >92%; or c) the LB of the 97.5%CI for the difference was above the non-inferiority margin of -6% and the LB of the 95%CI for the SVR12 rate within Arm C was below 92%; Difference in percentage of participants = -0.4, 95% CI 2-sided [-4.8 to 4.0]
Statistical Analysis 2: Comparison: Arm C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage of participants = 94.9, 97.5% CI 2-sided [91.0 to 98.8]
Statistical Analysis 3: Comparison: Arm A vs Arm C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage of participants = -0.4, 97.5% CI 2-sided [-5.4 to 4.6]

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12): Superiority of Arm A to Arm B
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug. Per statistical analysis plan to adjust for multiplicity among the primary and first secondary hypothesis tests, the test for superiority of Arm A to Arm B was not conducted.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 233 | 115
percentage of participants | 95.3 [92.6 to 98.0] | 96.5 [93.2 to 99.9]

4. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Time Frame: Treatment weeks 1, 2, 4, 8 (end of treatment for Arm C), and 12 (end of treatment for Arms A and B) or premature discontinuation from treatment
Population: All participants who received at least 1 dose of study drug (ITT population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 233 | 115 | 157
percentage of participants | 0.4 [0.1 to 2.4] | 0 [0.0 to 3.2] | 0.6 [0.1 to 3.5]

5. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment, excluding reinfection.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 222 | 114 | 150
percentage of participants | 1.4 [0.5 to 3.9] | 0.9 [0.2 to 4.8] | 3.3 [1.4 to 7.6]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Arm A | ARM B | ARM C
Serious Adverse Events (participants affected / at risk) | 5/233 | 2/115 | 3/157
Other Adverse Events (participants affected / at risk) | 126/233 | 53/115 | 64/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=233) | ARM B (N=115) | ARM C (N=157)
ULCERATIVE KERATITIS (Eye disorders) | 0 | 0 | 1
OPHTHALMIC HERPES SIMPLEX (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0
PARANASAL SINUS AND NASAL CAVITY MALIGNANT NEOPLASM RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
DEPENDENCE (Psychiatric disorders) | 0 | 0 | 1
SUBSTANCE-INDUCED PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=233) | ARM B (N=115) | ARM C (N=157)
DIARRHOEA (Gastrointestinal disorders) | 15 | 4 | 18
NAUSEA (Gastrointestinal disorders) | 32 | 15 | 19
VOMITING (Gastrointestinal disorders) | 10 | 5 | 9
ASTHENIA (General disorders) | 4 | 7 | 3
FATIGUE (General disorders) | 44 | 16 | 20
NASOPHARYNGITIS (Infections and infestations) | 12 | 6 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 15 | 4 | 2
HEADACHE (Nervous system disorders) | 60 | 21 | 31
INSOMNIA (Psychiatric disorders) | 9 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.